CLINICAL TRIAL: NCT04919915
Title: Home Air in Agriculture: Pediatric Intervention Trial
Acronym: HAPI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Environmental Health Sciences (NIEHS) (NIH); National Institute for Biomedical Imaging and Bioengineering (NIBIB) (NIH); The Yakima Valley Farm Workers Clinic (Other)
Responsible Party: Principal Investigator, Catherine Karr, Professor, School of Medicine: Pediatrics, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00001292; 5R01ES023510-03 (NIH); U01EB021923 (NIH); P30ES007033 (NIH); U2CES026561 (NIH)
Record Dates: First submitted 2021-05-19; First posted 2021-06-09 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-06

CONDITIONS: Asthma in Children
Keywords: Latinx children; agriculture; HEPA air cleaner; home indoor/outdoor sampling; coarse particulate matter; fine particulate matter; endotoxins; antigens; spirometry; exhaled nitric oxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Other): Households are randomly assigned to the intervention group with asthma education and received two HEPA air cleaners designed to reduce PM and NH3.
  Interventions: Device: HEPA air cleaner
- Control group (No Intervention): Households are randomly assigned to the control group. They only received the asthma education during the study period. These households receive a HEPA air cleaner at the end of the study.

INTERVENTIONS:
Device: HEPA air cleaner — Participants in the intervention group received two HEPA air cleaners per household. They were informed to place the HEPA air cleaners in the child's bedroom and the living room. Field staff provided and discuss how to use the air cleaner which promoted continuous operation of both air cleaners, keeping the child's bedroom door closed, and selected the highest fan speed. Typical use of the HEPA cleaners were questioned during the mid-study and final visits.
  Arms: Intervention group

SUMMARY:
This study seeks to reduce exposure to asthmagens in the homes of a community of Latino children residing in an area of intense agricultural production in Eastern Washington by testing the effectiveness of an intervention (high efficiency particulate air filter- HEPA portable room air cleaners) plus asthma education to reduce indoor measures of particulate matter, ammonia, improve clinically relevant measures of asthma health, and reduce biomarkers of inflammation.

DETAILED DESCRIPTION:
Over the course of five years, this project's specific aims are as follows:

1. Build on a well-established community based participatory research program to engage community partners in the design, implementation and evaluation of this asthma intervention study.
2. Conduct a year-long intervention study with longitudinal measurement of key asthmagen exposures and health outcome indicators with minimal participant burden.
3. Develop and characterize evaluation metrics for the process, impact and outcomes of this project in achievement of the aims.
4. Promote sustainable public health action via positive and transparent communications about the project to participants, local stakeholders, and state level policy makers through broad-based community outreach.

ELIGIBILITY:
Inclusion Criteria:

* Eligibility criteria include male and female, poorly controlled asthma, likely to stay in the area over the course of the study, having only one residence, no smokers in the household and residential proximity to dairy operations/crop production (<400 meters) determined by the telephone screening questionnaire.

Exclusion Criteria:

* Prior participation in the Asthma Home Visiting Program, not from the northern third of the lower Yakima Valley, well controlled asthma, unlikely to stay in the are over the course of the study, smokers in the household, no residential proximity to dairy operations or crop production, having more than one residence and inability to communicate over the phone.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 71 (Actual)
Dates: Start 2015-07-14 (Actual); Primary Completion 2019-02-27 (Actual); Study Completion 2019-02-27 (Actual)

PRIMARY OUTCOMES:
Change in particulate matter 2.5 (PM2.5) concentration | 1 year (study period)
  Indoor air sampling for PM2.5 collected over a 14-day period. MicroPEM (RTI International, Research Triangle Park, NC, USA) is turn on and left on for 14 days. Measurements collected at beginning and at 1 year after enrollment.
Change in ammonia (NH3) concentration | 1 year (study period)
  Indoor air sampling for NH3 collected over a 14-day period. Ogawa passive sampler (Ogawa USA, Pompano Beach, Fl, USA) is left open for 14 days. Measurements collected at beginning and at 1 year after enrollment.
Asthma Control Test | At study enrollment
  ACT score using the ACT questionnaire
Clinical utilization | One year (study period)
  Caregivers were asked if child had a scheduled or unscheduled ("urgent") clinical visit with a doctor or health care provider, emergency department, or overnight hospitalization for asthma symptoms. Number and types of visits are reported.
Inflammatory markers of asthma: Urinary leukotriene | 1 year (study period)
  Measured urinary leukotriene concentration and specific gravity in child urine sample. Measurements collected at enrollment, mid-study (4-6 months after enrollment), and end of study (1 year after enrollment)
Inflammatory markers of asthma: Fractional exhaled nitric oxide | At study enrollment
  Portable NIOX VERO (Aerocrine Inc, Stockholm, Sweden) for direct measurement of fractional exhaled nitric oxide.
Asthma exacerbation | One year (study period)
  Reviewed participant medical records for receipt of prescription for a course of oral corticosteroid.
Lung function | At study enrollment
  Measured lung fuction using EasyOne spirometer (NDD Technologies, Andover, MA). Minimum of three exhalations with acceptable starts, complete exhalation, and no coughs until two exhalations with acceptable repeatability was achieved.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Karr, MD, PhD, Principal Investigator — University of Washington
Locations (1):
- Yakima Valley Farmworkers Clinic, Yakima, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
Data has been shared with the NIH Chear Lab as part of U2CES02651
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Background] Masterson EE, Younglove LB, Perez A, Torres E, Krenz JE, Tchong French MI, Riederer AM, Sampson PD, Metwali N, Min E, Jansen KL, Aisenberg G, Babadi RS, Farquhar SA, Thorne PS, Karr CJ. The home air in agriculture pediatric intervention (HAPI) trial: Rationale and methods. Contemp Clin Trials. 2020 Sep;96:106085. doi: 10.1016/j.cct.2020.106085. Epub 2020 Jul 25. PMID 32721578
- [Background] Riederer AM, Krenz JE, Tchong-French MI, Torres E, Perez A, Younglove LR, Jansen KL, Hardie DC, Farquhar SA, Sampson PD, Karr CJ. Effectiveness of portable HEPA air cleaners on reducing indoor PM2.5 and NH3 in an agricultural cohort of children with asthma: A randomized intervention trial. Indoor Air. 2021 Mar;31(2):454-466. doi: 10.1111/ina.12753. Epub 2021 Jan 22. PMID 32996146
- [Derived] Drieling RL, Sampson PD, Krenz JE, Tchong French MI, Jansen KL, Massey AE, Farquhar SA, Min E, Perez A, Riederer AM, Torres E, Younglove LR, Aisenberg E, Andra SS, Kim-Schulze S, Karr CJ. Randomized trial of a portable HEPA air cleaner intervention to reduce asthma morbidity among Latino children in an agricultural community. Environ Health. 2022 Jan 3;21(1):1. doi: 10.1186/s12940-021-00816-w. PMID 34980119